CLINICAL TRIAL: NCT04573062
Title: Natural History of Post-Coronavirus Disease 19 Convalescence at the National Institutes of Health
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000089; 000089-N
Record Dates: First submitted 2020-10-01; First posted 2020-10-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10-07

CONDITIONS: Post-Coronavirus Disease 19
Keywords: Post-COVID-19; Convalescence; COVID-19; COVID; PASC; Natural History
MeSH Terms: conditions — Convalescence; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post COVID patients: Individuals whom have previously had COVID -19 infection.

SUMMARY:
Background:

People who get COVID-19 have a wide range of symptoms. They also recover from COVID-19 in different ways. In this study, researchers will use survey data to describe the different ways people experience and recover from COVID-19. They will also use the data to help create future studies to understand why some people do not fully recover.

Objective:

To learn more about the range and timing of symptoms that people have before, during, and after COVID-19 infection.

Eligibility:

People ages 18 and older who can give documentation of a positive COVID-19 or antibody test.

Design:

Participants will be screened with a telephone interview. It will take 15 minutes. They will provide their COVID-19 test results and medical records.

Participants will complete a second telephone interview. It will take 30 60 minutes. They will also take online surveys every 3 months for 3 years.

The interview and surveys will ask participants about their health before they got COVID-19, what happened while they had COVID-19, and what their recovery has been like.

Participants will get log-in data to take the online surveys. Completing all of the surveys the first time may take up to 3 hours. Follow-up surveys will take up to 30 minutes. Participants do not have to complete the surveys in one sitting. They will be able to save their progress and finish the surveys later.

Participants may be contacted to take part in other research studies.

DETAILED DESCRIPTION:
Study Description:

In late 2019, the novel coronavirus SARS/CoV2 appeared in Wuhan, China. The various ways that humans will recover from COVID-19 is just starting to be observed and it is clear there will be a wide range of convalescent experiences. A year into the pandemic, the post-acute sequelae of SARS/CoV2 infection (PASC) is known to be common and includes a broad range of symptoms and potential pathologies. This phased protocol is designed to observe and study the convalescence and recoveries from acute SARS/CoV2 infections.

Phase A Phase A Surveying (Phase A) will enable people in the community that are convalescing from COVID-19 to be studied using telephone interviews and internet-based questionnaires. The objective of Phase A Surveying is to observe and describe the range of medical syndromes that occur in the wake of an acute SARS/CoV2 infection.

Participants are required to be within the first five years of their recovery and have documentation of a positive laboratory test for COVID-19. Additional cohorts of persons with neurological sequelae, persons with a clinical diagnosis of COVID-19 with negative testing, persons with adverse complications after COVID 19 vaccination and participants co-enrolled in other research studies within the Division of Intramural Research will also be studied. The data collected during Phase A will describe the range of symptoms and patterns of symptom clustering of PASC. This data will also characterize the patient populations which have been or will be evaluated at the NIH Clinical Center in more detail.

Phase B Evaluation (Phase B) will allow surveyed participants of research interest from Phase A to be invited to the NIH Clinical Center for a medical evaluation and to undergo a panel of standard research measurements. Each participant will be medically and psychologically characterized to best understand if their complaints can be attributed to known disorders. The observations made during Phase B will provide insights into the range, character, and subtypes of PASC. Individuals found to have disorders being studied within the Division of Intermural Research at NIH will be appropriately referred.

Evaluated individuals with persistent symptoms in the absence of other demonstrable medical disease and individuals who fully recovered from a confirmed SARS/CoV2 infection will be invited back to the NIH Clinical Center for broad and deep research measurements.

Phase C Deep Phenotyping (Phase C) will be synchronized with other NIH-approved deep phenotyping protocols to foster cross-phenotype comparison research with other medical syndromes, such as Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) and Gulf War Illness (GWI). Deep phenotyping characterizations would be used to generate scientific hypotheses for testing in future studies and for cross-comparisons with other fatiguing disorders.

Previous epidemics have created unique medical syndromes in the past. Data from this protocol may be used to characterize PASC and any Post-COVID 19 Syndrome subtypes that may be discovered. If warranted, a Criteria Development phase will develop data-driven research consensus criteria for defining PASC and any Post-COVID 19 Syndromes.

The results of this protocol will provide novel insights into COVID-19 convalescence and its potential outcomes.

This current version of the protocol provides the details for Phase A, Phase B, and Phase C. Additional phases will be detailed in planned protocol amendments.

Objectives:

Primary Objective:

Phase A: To observe and describe the range of medical syndromes that occur in the wake of acute SARS/CoV2 infection.

Phase B: To describe and medically characterize patients with PASC and those who fully recovered from SARS/CoV2 infection.

Phase C: To compare the clinical and biological phenotypes between persons with unexplained PASC and those who fully recovered from SARS/CoV2 infection.

Secondary Objectives:

Phase A:

* To observe and describe recovery trajectories following an acute SARS/CoV2 infection.
* To observe and describe the range of medical syndromes and recovery trajectories of participants who report adverse effects after COVID-19 vaccination.
* To compare the range of medical syndromes and recovery trajectories of participants with a confirmed SARS/CoV2 infection to other cohorts, such as participants who have a medically confirmed diagnosis of COVID-19 without laboratory confirmation and participants who report adverse complications after COVID-19 vaccination.

Phase B:

* To determine the relations between acute SARS/CoV2 severity, subjective functional impairment, and objective functional performance.
* To explore the pathophysiology of PASC and its subtypes.

Phase C:

* To compare the clinical and biological phenotypes between persons with PASC to historic data and samples collected on persons with post-infectious Myalgic Encephalomyelitis/Chronic Fatigue Syndrome, and veterans with Gulf War Illness.
* To explore the pathophysiology of fatigue and post-exertional malaise in PASC. Fatigue will be explored using tasks designed to create muscular and cognitive fatigue. Post-exertional malaise will be explored using an exercise stress test and measuring the symptomatic and biological changes.

Endpoints:

Outcome measures

Phase A: The number and severity of persistent symptoms associated with COVID-19 convalescence. Collected data will be used to characterize different narratives of COVID-19 convalescence.

Phase B: Collected data and samples for use to perform exploratory analyses for the generation of new hypotheses regarding PASC.

Phase C: Identification of hypothetical mechanisms of PASC using collected data and samples. The types of analyses to be performed will be wide ranging. Planned exploratory areas of focus may include:

1. Immune system and inflammatory signaling characterization in at baseline and following maximal exercise exertion using flow cytometry, RNA sequencing, multiplex immunochemical analysis, NK cell functional analysis.
2. Microbiome characterization at baseline and following maximal exercise exertion using shotgun metagenomics.
3. Bioenergetics, autonomic, and metabolic characterization using mitochondrial plasmid genotyping, pulmonary spirometry, gas exchange measurements during exercise, metabolic chamber measurements of total body energy use, metabolomic analysis of stool, mitochondrion proteomics and metabolomics from muscle, and functional respiration of PBMCs using extracellular flux mito stress assay.
4. Characterization of physical and cognitive fatigue using functional magnetic resonance imaging and transcranial magnetic stimulation at baseline and following maximal exercise exertion.
5. Characterization of neurocognition at baseline and following maximal exercise exertion.

ELIGIBILITY:
* INCLUSION CRITERIA:

For Phase A Surveying:

1590 persons who are recovering or have recovered from an acute SARS/CoV2 infection will participate.

Inclusion criteria for Phase A:

Post-COVID-19 Convalescence (n=890)

1. Participants 18 and older
2. Ability to provide informed consent
3. Stated willingness to complete telephone interviews

4 Reports having begun recovery from an acute SARS/CoV2 infection in the past 5 years

a.For participants who don t have a known recovery date, a date of 6 weeks from infection will be imposed

5 Provides documentation of a positive COVID-19 Test. Approved test can include the following:

1. PCR, NAA, or other EUA Approved test to confirm active COVID infection.
2. A positive home Antigen test is acceptable when documentation of a photograph of the test with a phone-based date and time stamp is provided.
3. A positive anti-Spike antibody test is accepted in unvaccinated individuals or those who had antibody testing prior to vaccination.
4. A positive anti-nucleocapsid antibody test

   OR

   Test-Negative COVID-19 with Persistent Symptoms (n=50)
   1. Participants 18 and older
   2. Ability to provide informed consent
   3. Stated willingness to complete telephone interviews
   4. Reports having developed persistent symptoms as a consequence of an acute SARS/CoV2 infection
   5. Provides documentation of a clinical diagnosis of an acute SARS/CoV2 infection from a medical practitioner OR meets the Clinical Criteria of the 2020 CDC Interim Case Definition for Probable SARS/CoV2 infection.
   6. Has either negative or absent COVID-19 PCR, NAA, or other EUA Approved testing for the documented SARS/COV2 infection.
   7. Provides documentation of a negative COVID-19 antibody test prior to vaccination.

   OR

   COVID-19 vaccine related medical conditions (n=50)
   1. Participants 18 and older
   2. Ability to provide informed consent
   3. Stated willingness to complete telephone interviews
   4. Reports having developed persistent symptoms as a consequence of a COVID 19 vaccination
   5. Provides documentation of COVID-19 vaccination
   6. Provides documentation of a COVID-19 vaccine related medical condition from a medical practitioner

   OR

   Participants with a history of multiple SARS-CoV-2 infections (N=600)
   1. Participants 18 and older
   2. Ability to provide informed consent
   3. Stated willingness to complete telephone interviews
   4. Reports having more than one SARS-CoV-2 infection
   5. Provides documentation of at least one positive COVID-19 Test. Approved test can include the following:
5. PCR, NAA, or other EUA Approved test to confirm active COVID infection.
6. A positive home Antigen test is acceptable when documentation of a photograph of the test with a phone-based date and time stamp is provided.
7. A positive anti-Spike antibody test is accepted in unvaccinated individuals or those who had antibody testing prior to vaccination.
8. A positive anti-nucleocapsid antibody test

   The elements of the 2020 CDC Interim Case Definition for Probable COVID-19 used for this protocol will be the Clinical Criteria:

   Clinical Criteria:

   At least two of the following symptoms: fever (measured or subjective), chills, rigors, myalgia, headache, sore throat, new olfactory and taste disorder(s)

   OR

   At least one of the following symptoms: cough, shortness of breath, or difficulty breathing

   OR

   Severe respiratory illness with at least one of the following:
   * Clinical or radiographic evidence of pneumonia, OR
   * Acute respiratory distress syndrome (ARDS).

   AND

   No alternative more likely diagnosis

   For Phase B Evaluation:

   240 persons who are recovering or have recovered from COVID-19 within the last five years will participate. The accrual ceiling is 120 PASC and 120 healthy volunteers, with a goal to identify 80 PASC participants and 80 post-COVID fully recovered healthy volunteers who may be eligible for Phase C. Time since infection (i.e. within first six months, six months to one year, one year to two years, and two years to five years) will also be considered, with a goal of recruiting at least 20 PASC participants and 20 post- COVID fully recovered participants within each of these four time frames.

   Inclusion Criteria for all Phase B participants:
   1. Adult participants aged 18 years and older
   2. Self-reported completion of at least the 7th grade of school.
   3. Fluency in English.
   4. Willing and able to complete all study procedures
   5. Participant has a primary care provider at the time of enrollment.
   6. Able to provide informed consent
   7. Participants must be at least six weeks out since the onset of COVID-19 symptoms with no fever for at least one week.
   8. Participants must be within five years since starting to recover from acute COVID- 19 symptoms. The date of the start of recovery can be determined by:

      * The date that fever broke for the first time
      * The date the participant recalls starting to improve
      * If a participant is unable to report a reliable date, a date of six weeks from the onset of COVID-19 symptoms may be imputed.
   9. Does not have an active SARS-CoV-2 infection. The protocol will conform with NIH CC standards for documenting a participant does not have active SARS-CoV- 2 infection. This may include screening interviews and/or testing.

   Additional Inclusion Criteria for Mild to Moderate Illness COVID-19 with severe PASC symptoms:
   1. Licensed Independent Practitioner documentation of a stable state of general well- health and physical function prior to contracting SARS-CoV-2. This may include medical records, correspondence letters, or information gathered from telephone calls with study personnel.
   2. A self-reported illness narrative of the development of persistent PASC symptoms after recovering from a SARS-CoV-2 infection. These include symptoms such as fatigue, cognitive difficulties, orthostatic intolerance, unrefreshing sleep, neuropathic pain, mood change, and post-exertional malaise.
   3. Laboratory documentation of a positive COVID-19 PCR, NAA, or other EUA Approved test to confirm active COVID infection at the time of the SARS-CoV-2 infection. Participants with positive home tests during Phase A will be required to have a positive anti-SARS nucleocapsid antibody test.
   4. Meets WHO Clinical Progression Scale of 2 - 6:

      * 2: Ambulatory; symptomatic, independent
      * 3: Ambulatory; symptomatic, assistance needed
      * 4: Hospitalized; no oxygen therapy
      * 5: Hospitalized; oxygen by mask or nasal prongs
      * 6: Hospitalized; oxygen by non-invasive ventilation or high flow oxygen
   5. Functional Criteria: Substantial symptom severity as determined using SF-36v2: score of <=70 physical function subscale, or <=50 on role physical subscale, or <=75 on social function subscale.

   OR

   Additional Inclusion Criteria for Mild or Moderate Illness COVID-19 without PASC symptoms:
   1. Licensed Independent Practitioner documentation of a stable state of general well- health and physical function prior to contracting SARS-CoV-2. This may include medical records, correspondence letters, or information gathered from telephone calls with study personnel.
   2. A self-reported illness narrative of recovery to prior health after a SARS/CoV2 infection.
   3. Laboratory documentation of a positive COVID-19 PCR, NAA, or other EUA Approved test to confirm active COVID infection at the time of the SARS-CoV-2 infection. Participants with positive home tests during Phase A will be required to have a positive anti-SARS nucleocapsid antibody test.
   4. Meets WHO Clinical Progression Scale of 2 - 6:

      * 2: Ambulatory; symptomatic, independent
      * 3: Ambulatory; symptomatic, assistance needed
      * 4: Hospitalized; no oxygen therapy
      * 5: Hospitalized; oxygen by mask or nasal prongs
      * 6: Hospitalized; oxygen by non-invasive ventilation or high flow oxygen

   Functional Criteria: No substantial symptom severity as determined using SF-36v2: score of >=85 physical function subscale, and >= 85 on role physical subscale, and >= 85 on social function subscale.

   OR

   Additional Inclusion Criteria for Mild or Moderate Illness COVID-19 with mild to moderate PASC symptoms:
   1. Licensed Independent Practitioner documentation of a stable state of general well-health and physical function prior to contracting SARS-CoV-2. This may include medical records, correspondence letters, or information gathered from telephone calls with study personnel.
   2. Either a self-reported illness narrative of near recovery to prior health or a narrative of the development of persistent PASC symptoms after recovering from a SARS-CoV-2 infection. These include symptoms such as fatigue, cognitive difficulties, orthostatic intolerance, unrefreshing sleep, neuropathic pain, mood change, and post-exertional malaise.
   3. Laboratory documentation of a positive COVID-19 PCR, NAA, or other EUA Approved test to confirm active COVID infection at the time of the SARS-CoV-2 infection. Participants with positive home tests during Phase A will be required to have a positive Anti-SARS nucleocapsid antibody test.
   4. Meets WHO Clinical Progression Scale of 2 - 6:

      * 2: Ambulatory; symptomatic, independent
      * 3: Ambulatory; symptomatic, assistance needed
      * 4: Hospitalized; no oxygen therapy
      * 5: Hospitalized; oxygen by mask or nasal prongs
      * 6: Hospitalized; oxygen by non-invasive ventilation or high flow oxygen
   5. Functional Criteria: Mild to moderate symptom severity as determined using SF-36v2: score of between 71 and 84 on the physical function subscale, or between 51 and 84 on role physical subscale, or between 76 and 84 on social function subscale.

   For Phase C Deep Phenotyping:

   Inclusion Criteria for Mild to Moderate Illness COVID-19 with PASC symptoms:
   1. Met inclusion and exclusion criteria for Mild to Moderate Illness COVID-19 with severe post-acute COVID-19 symptoms after completing Phase B.
   2. No alternative explanation for PASC symptoms identified by adjudication committee during Phase B.
   3. Fluency in English

   OR

   Inclusion Criteria for Mild or Moderate Illness COVID-19 without PASC symptoms:
   1. Met inclusion and exclusion criteria for Mild to Moderate Illness COVID-19 without post-acute COVID-19 symptoms after completing Phase B.
   2. Fluency in English

   EXCLUSION CRITERIA:

   Exclusion criteria for Phase A:
   1. Not willing to provide personal identifying information to investigative team
   2. Cognitive impairment that is severe enough to limit consent capacity

   Exclusion criteria for Phase B Evaluation:

   Information collected from Phase A interviews, review of medical records, and discussions with consented Phase A participants will be used to determine if a participant will be excluded from participation.
   1. Current or past psychotic disorder including depression with psychosis, bipolar disorder with psychotic symptoms and schizophrenia
   2. Major depression disorder, generalized anxiety disorder, post-traumatic stress disorder, panic disorder, or obsessive-compulsive disorder unless managed for more than six months with a stable treatment regimen
   3. Current or past substance use disorder within last five years. Marijuana use within the past five years will not be an exclusion.
   4. Positive urine toxicology screening for anything other than marijuana. Positive result for corresponding medication prescribed for short-term medical issue may be allowed after investigator review. Examples include use of a benzodiazepine prior to air travel to NIH or narcotic medication related to a recent medical procedure or injury.
   5. Current suicidal ideation
   6. History of head injury leading to moderate or severe traumatic brain injury. Persons having a history of mild TBI (mTBI) will not be excluded.
   7. Women who are pregnant, breastfeeding, or are within one-year post-partum.
   8. Current or previous malignancy. A history of malignancy that has fully resolved with surgical resection only (e.g. no chemotherapy, radiation therapy, or immunotherapy) will be allowed.
   9. Current systemic immunologic disorders (e.g. Type 1 diabetes, rheumatoid arthritis). Local immunological disorder (e.g. atopic dermatitis, stable autoimmune thyroid disease) and allergic disorders will be allowed.
   10. Current or previous long-term immune suppressive therapy. Recent or current steroid use for the treatment of COVID-19, PASC, recent allergic reactions, and topical steroid use is allowed.
   11. Any premorbid medical condition that would potentially cause fatigue and exercise intolerance that would exclude from participation in Phase C. This includes many chronic medical diseases, such

       as congestive heart failure, coronary artery disease, chronic obstructive pulmonary disease, severe arthritis, uncontrolled asthma, renal failure, fibromyalgia, and ME/CFS.
   12. Active participation in a clinical protocol (e.g. anti-inflammatory drug intervention study) which includes an intervention that may affect the results of the current study.
   13. Not willing to allow for research data and samples to be shared broadly with other researchers.
   14. Employees at NIH that are under the direct supervision of the study investigators (family members of NIH employees are permitted to participate).
   15. Symptom severity that makes it impossible for the volunteer to travel to NIH.

   Exclusion criteria for Phase C Deep Phenotyping:

   Exclusion criteria for all Phase C participants:
   1. Current or past psychotic disorder including depression with psychosis, bipolar disorder with psychotic symptoms and schizophrenia
   2. Current DSM-5-defined major depression disorder, generalized anxiety disorder, post-traumatic stress disorder,...

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1590 persons within five years of convalescence of a single acute SARS-CoV-2 will participate, including at least 250 adults recovering from neurological sequelae. Additional cohorts of 50 adults with a clinical diagnosis of SARS-CoV-2 infection with negative or absent PCR testing and negative antibody testing and 50 adults with medical documentation of a COVID-19 vaccine related medical condition will be enrolled. Participants in NIH protocols 20CC0113: Cardiopulmonary Inflammation and Multi-System Imaging During the Clinical Course of COVID-19 Infection in Asymptomatic and Symptomatic Persons and 000102-CC: COVID-19, Chronic Adaptation, and Response to Exercise may also co-enroll. Up to 240 Phase A participants will complete a Phase B research evaluation. Additionally, 80 unexplained PASC participants and 80 post-COVID recovered controls who completed Phase B will be invited for a Phase C deep phenotyping visit, with a target of completing measures on 50 in each group.
Sampling Method: Non-Probability Sample
Enrollment: 1590 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Screening Phase | End of Study
  The number and severity of persistent symptoms associated with COVID-19 convalescence. Collected data will be used to characterize different narratives of COVID-19 convalescence.
Phase C: Deep Phenotyping | End of Study
  Phase C: Immune system and inflammatory signaling characterization in at baseline and following maximal exercise exertion using flow cytometry, RNA sequencing, multiplex immunochemical analysis, NK cell functional analysis. Microbiome characterization at baseline and following maximal exercise exertion using shotgun metagenomics. Bioenergetics, autonomic, and metabolic characterization using mitochondrial plasmid genotyping, pulmonary spirometry, gas exchange measurements during exercise, metabolic chamber measurements of total body energy use, metabolomic analysis of stool, mitochondrion proteomics and metabolomics from muscle, and functional respiration of PBMCs using extracellular flux mito stress assay.
Phase B: Evaluation | End of Study
  Phase B: Standard clinical and research evaluations will be used to measure cardiopulmonary, neurological, and functional status and identify individuals with unknown PASC.

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Walitt, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pan L, Mu M, Yang P, Sun Y, Wang R, Yan J, Li P, Hu B, Wang J, Hu C, Jin Y, Niu X, Ping R, Du Y, Li T, Xu G, Hu Q, Tu L. Clinical Characteristics of COVID-19 Patients With Digestive Symptoms in Hubei, China: A Descriptive, Cross-Sectional, Multicenter Study. Am J Gastroenterol. 2020 May;115(5):766-773. doi: 10.14309/ajg.0000000000000620. PMID 32287140
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Chen ATC, Coura-Filho GB, Rehder MHH. Clinical Characteristics of Covid-19 in China. N Engl J Med. 2020 May 7;382(19):1860. doi: 10.1056/NEJMc2005203. Epub 2020 Mar 27. No abstract available. PMID 32220203
- [Derived] Huff HV, Roberts H, Bartrum E, Norato G, Grayson N, Fleig K, Wilkerson MJ, Stussman BJ, Nath A, Walitt B. Prevalence and severity of neurologic symptoms in Long-COVID and the role of pre-existing conditions, hospitalization, and mental health. Front Neurol. 2025 Jun 25;16:1562084. doi: 10.3389/fneur.2025.1562084. eCollection 2025. PMID 40635708
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000089-N.html